CLINICAL TRIAL: NCT04149392
Title: Pilot Study for the Use of CGM for Post-discharge Diabetes Management Following a Hospitalization for Heart Failure or MI
Brief Title: Use of CGM for Diabetes Management Following a Hospitalization.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Changed to quality improvement project
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Heather Ferris, Physician scientist, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15055
Record Dates: First submitted 2019-10-29; First posted 2019-11-04 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Diabetes
Keywords: CGM Diabetes Heart Failure
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CGM intervention (Experimental): Patients with diabetes hospitalized for heart failure or acute myocardial infarction will have a continuous glucose monitor (CGM) placed on the day of discharge which will be downloaded at their outpatient follow up clinic visit 6-14 days later. At the follow-up visit medications may be modified based on downloaded glucose data. During the already scheduled post-discharge follow up appointment the CGM sensor data will be downloaded by clinic staff. The diabetes medications will be reconciled and the downloaded data will be reviewed with the patient. Based on the download, a PharmD will have the option of increasing or decreasing insulin doses by a maximum of 10% to reduce hypoglycemia and/or hyperglycemia. The goal will be to adjust medications, if needed, to target blood sugars between 90-250mg/dl greater than 80% of the time.
  Interventions: Device: Continuous Glucose Monitor

INTERVENTIONS:
Device: Continuous Glucose Monitor — Patients with diabetes hospitalized for heart failure or acute myocardial infarction will have a continuous glucose monitor (CGM) placed on the day of discharge. The participants will go home with the device and keep it for 6-14 days until they return to clinic for follow up visit. At this time the device will be removed, the information regarding glucose levels during those days will be downloaded and based on the download, a PharmD will have the option of increasing or decreasing insulin doses by a maximum of 10% to reduce hypoglycemia and/or hyperglycemia. The goal will be to adjust medications, if needed, to target blood sugars between 90-250mg/dl greater than 80% of the time.

SUMMARY:
Patients with diabetes hospitalized for heart failure or acute myocardial infarction will have a continuous glucose monitor (CGM) placed on the day of discharge which will be downloaded at their outpatient follow up clinic visit 6-14 days later. At the follow-up visit medications may be modified based on downloaded glucose data. This study is designed to determine the frequency that patients with diabetes hospitalized for heart failure or acute myocardial infarction have significant hypoglycemia or hyperglycemia requiring medication adjustment in the 1-2 weeks following hospital discharge. The outcome will be a binary- yes, diabetes medications were adjusted or no, diabetes medications were not adjusted.

As a secondary outcome 30-day hospital readmission and mortality will be compared to historical hospital data collected by the inpatient cardiovascular service as part of their quality improvement monitoring. Researchers do not expect to see a significant difference in 30-day readmission or mortality as this study will be under-powered. In addition, our inclusion criteria will specifically target the patients at highest risk for bad diabetes outcomes, thus researchers may see worse outcomes compared to historical controls, but this assessment will help us design future randomized studies.

DETAILED DESCRIPTION:
After the participant has signed the consent form a continuous glucose monitor (CGM) sensor will be placed on the arm of the participant. If consent is signed prior to the day of discharge the sensor placement will be delayed until the day of discharge. The participant will be provided with instruction to avoid bumping the sensor and to avoid dislodging when bathing and dressing. If the sensor should fall off before the follow up appointment, they will be instructed to bring it with them for a partial download.

During the already scheduled post-discharge follow up appointment the CGM sensor data will be downloaded by clinic staff. The diabetes medications will be reconciled, and the downloaded data will be reviewed with the patient. Based on the download, a PharmD will have the option of increasing or decreasing insulin doses by a maximum of 10% to reduce hypoglycemia and/or hyperglycemia. The goal will be to adjust medications, if needed, to target blood sugars between 90-250mg/dl greater than 80% of the time. This is a conservative goal aimed at reducing risk for severe hypo or hyperglycemia with good glycemic control rather than to target tight glycemic control. If adjustment of oral agents or a change of greater than 10% is required this will be done in consultation with an attending physician.

These adjustments will follow standards of care and the expectation is that this will benefit the patient. All changes will be communicated to the participant's primary care physician (PCP) or endocrinologist. If the patient does not have an endocrinologist and it is felt that significant adjustments will be required over time to improve the participant's glucose control they will be given the option of a referral to the Diabetes Cardiovascular Clinic, General Endocrinology Clinic, or if having excessive hypoglycemia the Diabetes Technology Clinic for consideration for long term use of CGM. If no changes are required, this will also be communicated to the patient's PCP or endocrinologist. The downloaded data from the CGM will be scanned in the media tab in the electronic medical record and any adjustments will be included as part of the medical record.

Between 30 and 40 days post-discharge the participant's medical record will be accessed again. At this point it will be determined if the patient was readmitted to the hospital or died in the 30 days post-discharge. In addition, clinic notes will be examined to determine if there is any evidence that the patient developed worsening hypoglycemia or worsening hyperglycemia in response to medication adjustments made during the post-discharge clinic. This data will be collected to assist in understanding the efficacy of the intervention and to ensure that the intervention is not causing unintended harm. This access of the medical record would not be expected to benefit the patient but could provide benefit to future participants or patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-100 years.
* Admitted to either the heart failure or acute coronary service.
* Followed by the cardiovascular diabetes service for at least 1 day during hospital admission.
* Planned follow up in either the UVA heart failure readmission clinic or the ACS readmission clinic in 6-14 days post-discharge.
* Use of insulin, a sulfonylurea, or evidence of poor diabetes control prior to admission.

Exclusion Criteria:

* Non-English speaking.
* Pregnant.
* Requiring dialysis.
* Lymphedema of both arms.
* Current CGM use.
* Plan for CT-scan, MRI or diathermy treatment within 14 days of discharge.
* Patients taking high dose vitamin C supplements (multivitamin is ok).
* Patients taking more than 325mg of aspirin daily.
* Discharge to skilled nursing facility or acute rehab.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-16 (Estimated); Primary Completion 2020-04-06 (Estimated); Study Completion 2020-04-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of diabetes medication changes that take place at the follow up visit | this will happen between the time of enrollment and the follow up clinic visit 6-14 days after enrollment.
  We will determine the frequency of diabetes medication changes that take place at the follow up visit.

SECONDARY OUTCOMES:
30-day Readmission rate | 30 days after hospital discharged
  Researchers will determine the 30-day readmission rate for participants.
Mortality rate | 30-40 days after hospital discharged
  Researchers will determine the mortality rate for participants.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Ferris, MD PhD, Principal Investigator — University of Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dungan K, Graessle K, Sagrilla C. The effect of congestive heart failure on sensor accuracy among hospitalized patients with type 2 diabetes. Diabetes Technol Ther. 2013 Oct;15(10):817-24. doi: 10.1089/dia.2013.0094. PMID 24050738
- [Background] Tung YC, Chang GM, Chang HY, Yu TH. Relationship between Early Physician Follow-Up and 30-Day Readmission after Acute Myocardial Infarction and Heart Failure. PLoS One. 2017 Jan 27;12(1):e0170061. doi: 10.1371/journal.pone.0170061. eCollection 2017. PMID 28129332
- [Background] Dei Cas A, Khan SS, Butler J, Mentz RJ, Bonow RO, Avogaro A, Tschoepe D, Doehner W, Greene SJ, Senni M, Gheorghiade M, Fonarow GC. Impact of diabetes on epidemiology, treatment, and outcomes of patients with heart failure. JACC Heart Fail. 2015 Feb;3(2):136-45. doi: 10.1016/j.jchf.2014.08.004. PMID 25660838
- [Background] Ruppar TM, Cooper PS, Mehr DR, Delgado JM, Dunbar-Jacob JM. Medication Adherence Interventions Improve Heart Failure Mortality and Readmission Rates: Systematic Review and Meta-Analysis of Controlled Trials. J Am Heart Assoc. 2016 Jun 17;5(6):e002606. doi: 10.1161/JAHA.115.002606. PMID 27317347
- [Background] Bergethon KE, Ju C, DeVore AD, Hardy NC, Fonarow GC, Yancy CW, Heidenreich PA, Bhatt DL, Peterson ED, Hernandez AF. Trends in 30-Day Readmission Rates for Patients Hospitalized With Heart Failure: Findings From the Get With The Guidelines-Heart Failure Registry. Circ Heart Fail. 2016 Jun;9(6):10.1161/CIRCHEARTFAILURE.115.002594 e002594. doi: 10.1161/CIRCHEARTFAILURE.115.002594. PMID 27301467
- [Background] Bilchick K, Moss T, Welch T, Levy W, Stukenborg G, Lawlor BT, Reigle J, Thomas SC, Brady C, Bergin JD, Kennedy JLW, Abuannadi M, Scully K, Mazimba S. Improving Heart Failure Readmission Costs and Outcomes With a Hospital-to-Home Readmission Intervention Program. Am J Med Qual. 2019 Mar/Apr;34(2):127-135. doi: 10.1177/1062860618788436. Epub 2018 Jul 19. PMID 30024279